CLINICAL TRIAL: NCT01825668
Title: Effect of a Plant Sterol-Fortified Low-fat Milk Product on Plasma Lipid Levels of Humans in Relation to Different Infant Feeding Practices and Later Life Cholesterol Metabolism
Brief Title: Effect of Plant Sterol Enriched Milk on Plasma Lipid Levels of Humans Breast-fed During Infancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B2013:019
Record Dates: First submitted 2013-03-21; First posted 2013-04-08 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2013-03

CONDITIONS: Hypercholesterolemia; CVD
MeSH Terms: conditions — Hypercholesterolemia | interventions — Phytosterols; Cholesterol, HDL

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High cholesterol (Experimental): 600 mg cholesterol/day in 240 ml milk shake
  Interventions: Other: High cholesterol
- Plant sterols (Experimental): 2.0 g of plant sterols/day in 240 ml milk shake containing 50 mg cholesterol
  Interventions: Other: Plant Sterols
- Placebo (Placebo Comparator): 50 mg cholesterol/day in 240 ml of milk shake
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Plant Sterols
  Arms: Plant sterols
Other: High cholesterol
  Arms: High cholesterol
Other: Placebo
  Arms: Placebo

SUMMARY:
The overall goal of this clinical study is to investigate how dietary cholesterol intake influences the plasma Total cholesterol (TC), LDL-Cholesterol levels and cholesterol metabolism between adults who had been breast-fed as infants as a function of the duration of breast feeding and quantity of early cholesterol intake. The study also aims to evaluate the effect of a plant sterol formulation in low fat milk shake in modulating the lipid profile favorably in the study population.

DETAILED DESCRIPTION:
Hypothesis 1: To determine the responsiveness of plasma lipid profile including Total cholesterol and LDL cholesterol concentrations to high and low cholesterol diets in adults who been breast-fed as infants for different durations

Hypothesis 2: To determine if differences exist in rates of cholesterol absorption and synthesis in adults, and whether such differences respond to variations in cholesterol intake, between individuals who were breast for different durations.

Hypothesis 3: Consumption of a plant sterol formulation in low-fat milk product will favorably alter lipid profiles compared with control in the study population.

This is a free-living, randomized, crossover trial. This trial is modeled after previously successful functional food trial at the investigators clinic, consistent with current recommendations to decrease Cardiovascular diseases (CVD) risk and improve circulating lipid profiles. The proposed study will include three treatment phases of 4 weeks each, separated by 4-week washout intervals:

Phase 1: Study diets with placebo (240 ml of 2% milk shake; 50 mg cholesterol).

Phase 2: Study diets with enriched cholesterol (240ml of 2% milk shake; 600 mg cholesterol).

Phase 3: A study diet with plant sterols (240 ml of 2% milk shake;2.0 g/d of plant sterols/240 ml serving; 50 mg cholesterol).

During each treatment period participants will consume their supper time meal along with assigned test product. Consumption of the suppertime meals and the test products will be monitored by a clinical coordinator to ensure compliance. Participants will be asked to fill out a 3-day food diary at the beginning and end of each experimental period.

ELIGIBILITY:
Inclusion Criteria:

* Triglycerides (TG) <3.0 mmol/L
* Body mass index (BMI) between 20 and 30 kg/m2
* Participants must have been breast-fed at least during the first 6 months of their life

Exclusion Criteria:

* History of recent (i.e. less than 1 month) or chronic use of oral hypolipidemic therapy, including fish oils, or probucol within the last 3 months
* History of chronic use of alcohol (>2 drinks/d), smoking, systemic antibodies, corticosteroids, androgens, or phenytoin
* Myocardial infarction, coronary artery bypass, kidney disease, liver disease or other major surgical procedures within the last six months,
* Sitosterolemic patients
* Recent onset of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, diabetes, or significant current (i.e. onset within past three months) gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year)
* Exercise greater than walking or running 15 miles/wk or 4,000 kcal/wk
* Participants who have not been breast-fed at all
* Pregnant or planning for pregnancy during the next 5 month period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in LDL-cholesterol | Day 1,2 & 29,30 of each of the 3 phases. Each phase duration is 1 month

SECONDARY OUTCOMES:
Change in Cholesterol Absorption | Day 26-30 of each of the 3 phases. Each phase duration is 1 month
  On day 26 of each dietary phase,a 12-hr fasting blood sample will be obtained to represent stable isotope baseline, after which participants will ingest 75 mg of the stable carbon isotope [3,4-13C] cholesterol stable isotope (13C-cholesterol)dissolved in 5 g of margarine and spread on half of an English muffin. Fasting blood samples will be taken also on days 27, 28, and 29 to monitor isotopic enrichment/decay levels. Free cholesterol extracted from the Red Blood Cell (RBC) fraction of blood will be used to determine 13C-cholesterol enrichment using on-line gas chromatography (GC)/combustion/isotope ratio mass spectrometry (IRMS)using previously established methods. Carbon-di-oxide (CO2) gas will be analyzed for 13C cholesterol enrichment against the Pee Dee Belemnite (PDB). From 24 to 96 hr, cholesterol absorption will be presented as area under the 13C cholesterol RBC enrichment curve calculated by the Number cruncher statistical system (NCSS) statistical software.
Change in Cholesterol Synthesis | Day 26-30 of each of the 3 phases. Each phase duration is 1 month
  On day 29 prior to breakfast, participants will consume 0.7 g/kg estimated body water (estimated at 60% of total body weight) of deuterium oxide (2H) as a tracer to measure cholesterol synthesis. Fasting blood sample will be collected after 24 hr (96 h after initial isotope administration) in order to monitor the change in deuterium enrichment within red blood cell (RBC) free cholesterol as an index of cholesterol synthesis.Free cholesterol will be extracted from RBC and water from plasma will be isolated using the blood samples collected from day 26-30 each phase. Cholesterol deuterium enrichment will be determined through being expressed relative to a series of standards using a GC/pyrolysis/IRMS using previously established methods. Cholesterol fractional synthesis rate (FSR) (% per day)will be calculated as the rate of incorporation of deuterium within the body water pool into RBC cholesterol pools by measuring the deuterium RBC enrichment over 24 hr.

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada